CLINICAL TRIAL: NCT02239965
Title: Qualitative Analysis of Barriers to Consistent Use of Neuromuscular Monitoring in General Anaesthesia
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jakob Louis Thomsen, MD, PhD student, Herlev Hospital
Other Study IDs: JLT-NM3
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade; Neuromuscular monitoring; Focus group interview; Clinical observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Anaesthesia personnel: Anaesthesiologists and nurse anaesthetists

SUMMARY:
Monitoring the degree of neuromuscular blockade in general anaesthesia reduces complications and patient discomfort. However, monitoring is not applied consistently by Danish anaesthesia personnel. Surveys show that part of the explanation is that the anaesthetists often experience problems with the equipment used for monitoring, though the problems have not been described in detail.

We hypothesise that the lack of consistent monitoring in general anaesthesia is caused by insecurity in the anaesthesia personnel's set-up and use of the equipment, as well as in interpreting the measurement results.

ELIGIBILITY:
Inclusion Criteria:

* has been working in the field of anaesthesiology for at least 1 year.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anaesthesiologists and nurse anaesthetists at Danish anaesthesia departments.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Description of the barriers to consistent neuromuscular monitoring, based on a qualitative analysis of focus group interviews with anaesthesiologists and nurse anaesthetists | Focus group interviews conducted Sep. - Oct. 2014 (2 months)
  Focus group interviews will collect participants' perspectives and will be analyzed for thoughts, opinions, and feelings in regard to neuromuscular monitoring. Specific problems experienced with the equipment and other possible barriers to the consistent use of monitoring will be described qualitatively.

SECONDARY OUTCOMES:
Description of the problems experienced with neuromuscular monitoring in daily clinical practice | Clinical observations conducted in Sep. - Oct. 2014 (2 months)
  The problems experienced with neuromuscular monitoring will be described through a qualitative analysis of clinical observations of the personnel's daily use of the monitoring equipment,

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark